CLINICAL TRIAL: NCT05667428
Title: A Multicenter Open-label Clinical Study on the Prevention of Premature Ovarian Failure After Hematopoietic Stem Cell Transplantation
Brief Title: A Multicenter Open-label Clinical Study on the Prevention of Premature Ovarian Failure After HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJTU1AF-CRF-2022-XK002
Record Dates: First submitted 2022-10-27; First posted 2022-12-28 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-10

CONDITIONS: Hematopoietic Stem Cell Transplantation; Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Leuprolide; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leprorelin group (Experimental): Leprorelin was given subcutaneously before each cycle of chemotherapy.
  Interventions: Drug: leuprorelin
- Control group (Placebo Comparator): Normal salinewas given subcutaneously before each cycle of chemotherapy.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: leuprorelin — From the initial chemotherapy after diagnosis, patients received a subcutaneous injection of leprorelin in each cycle of chemotherapy including the conditioning treatment prior to transplantation.
  Other Names: GnRHa
  Arms: Leprorelin group
Drug: normal saline — From the initial chemotherapy after diagnosis, patients received a subcutaneous injection of normal saline in each cycle of chemotherapy including the conditioning treatment prior to transplantation.
  Other Names: NS
  Arms: Control group

SUMMARY:
HSCT is an effective method to cure hematologic malignancies. However, the reproductive system is prone to be damaged during radiotherapy and chemotherapy before transplantation, leading to ovarian failure, followed by infertility and premature ovarian failure (POF), which seriously affect the long-term quality of life of patients. This clinical trial aimed to observe the effect of Gonadotropin-releasing hormone analogues (GnRHa) on ovarian function in women of reproductive age after HSCT, so as to provide clinical evidence for whether GnRHa should be used for the prevention of POF.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is an effective method for the treatment of hematologic malignancies. However, in the process of radiotherapy and chemotherapy before transplantation, the reproductive system is vulnerable to damage, leading to ovarian failure, which leads to infertility and premature ovarian failure (POF), seriously affecting the long-term quality of life of patients. Exogenous injection of gonadotropin-releasing hormone analogue (GnRHa) has a significant effect on fertility preservation in adolescent and reproductive female patients with breast cancer and cervical cancer. However, there is a lack of large-scale clinical studies on POF in HSCT. Therefore, this clinical trial aimed to observe the effect of GnRHa application before transplantation on ovarian function in women of reproductive age after transplantation, so as to provide clinical evidence for whether GnRHa application for fertility function protection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute leukemia, MDS, lymphoma, multiple myeloma, SAA and other hematological diseases, with the indications for autologous or allogeneic hematopoietic stem cell transplantation.
* Female, aged 18-45 years.
* Ovarian function was normal before treatment.
* Volunteer to participate in clinical research and sign the informed consent form.

Exclusion Criteria:

* No menstruation before treatment, undergone hysterectomy or ovarian surgery.
* Abnormal sexual development.
* Received radiotherapy.
* Combined with tumors affecting gonadal function.
* Deep vein thrombosis.
* Hypertension, liver and/or kidney dysfunction cannot tolerate hematopoietic stem cell transplantation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
POF rate | three years after transplantation
  Incidence of premature ovarian failure after transplantation

SECONDARY OUTCOMES:
acute GVHD rate | At day 100 post-transplantation
  the incidence of acute graft-versus-host disease (GVHD)
chronic GVHD rate | From date of HSCT until the end of follow-up or the date of death from any cause, whichever came first,assessed up to 36 months.
  the incidence of chronic graft-versus-host disease (GVHD)
PFS | From date of HSCT until the end of follow-up or the date of death from any cause, whichever came first，assessed up to 36 months.
  Progression Free Survival
OS | From date of diagnosis until the end of follow-up or the date of death from any cause, whichever came first，assessed up to 36 months.
  Overall Survival
AEs | up to 6 months after HSCT
  Adverse reations include abnormalities in bone mineral density, blood glucose, liver and kidney functions.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Wang, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China